CLINICAL TRIAL: NCT01939184
Title: A Study to Assess the Safety and Efficacy of WC3055 in Men With Lower Urinary Tract Symptoms (LUTS) Secondary to Benign Prostatic Hyperplasia (BPH)
Brief Title: Assess Safety & Efficacy of WC3055 in Men With Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR-05710
Record Dates: First submitted 2013-09-04; First posted 2013-09-11 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- WC3055-01F (Experimental): WC3055 12.5 mg tablet once daily for 12 weeks
  Interventions: Drug: WC3055
- WC3055-02F (Experimental): WC3055 25 mg tablet once daily for 12 weeks
  Interventions: Drug: WC3055
- WC3055-03F (Experimental): WC3055 50 mg tablet once daily for 12 weeks
  Interventions: Drug: WC3055
- WC3055-04F (Experimental): WC3055 75 mg tablet once daily for 12 weeks
  Interventions: Drug: WC3055
- WC3055-07P (Placebo Comparator): Placebo tablet once daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: WC3055 — 12.5, 25, 50 or 75 mg dose
  Arms: WC3055-01F; WC3055-02F; WC3055-03F; WC3055-04F
Other: Placebo — Placebo
  Arms: WC3055-07P

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of various fixed daily doses of WC3055 compared with placebo for the treatment of subjects with LUTS secondary to BPH.

ELIGIBILITY:
Inclusion Criteria:

* History of LUTS for ≥6 months secondary to BPH
* Total IPSS (International Prostate Symptom Score) ≥ 13 at Screening

Exclusion Criteria:

-

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Total IPSS (International Prostate Symptom Score) | Final Visit (Week 12 or final visit)
  Sum of Questions 1-7.

SECONDARY OUTCOMES:
Change from Baseline Total IPSS | Week 4
  Sum of Questions 1-7.
Change from Baseline Total IPSS | Week 8
  Sum of Questions 1-7.
Change from Baseline IIEF-EF (International Index of Erectile Function-Erectile Function) Domain Score | Week 4
  Questions 1, 2, 3, 4, 5, & 15.
Change from Baseline IIEF-EF Domain Score | Week 8
  Questions 1, 2, 3, 4, 5, & 15.
Change from Baseline IIEF-EF Domain Score | Week 12
  Questions 1, 2, 3, 4, 5, & 15.
Change from Baseline IIEF-EF Domain Score | Final Visit (Week 12 or Final Visit)
  Questions 1, 2, 3, 4, 5, & 15.

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Warner Chilcott
Locations (84):
- United States (84):
  - Warner Chilcott Investigational Study Site, Homewood, Alabama
  - Warner Chilcott Investigational Study Site, Huntsville, Alabama
  - Warner Chilcott Investigational Study Site, Mobile, Alabama
  - Warner Chilcott Investigational Study Site, Chandler, Arizona
  - Warner Chilcott Investigational Study Site, Gilbert, Arizona
  - Warner Chilcott Investigational Study Site, Glendale, Arizona
  - Warner Chilcott Investigational Study Site, Phoenix, Arizona
  - Warner Chilcott Investigational Study Site, Laguna Hills, California
  - Warner Chilcott Investigational Study Site, Murrieta, California
  - Warner Chilcott Investigational Study Site, San Diego, California
  - Warner Chilcott Investigational Study Site, Colorado Springs, Colorado
  - Warner Chilcott Investigational Study Site, Denver, Colorado
  - Warner Chilcott Investigational Study Site, Englewood, Colorado
  - Warner Chilcott Investigational Study Site, Parker, Colorado
  - Warner Chilcott Investigational Study Site, Middlebury, Connecticut
  - Warner Chilcott Investigational Study Site, New Britain, Connecticut
  - Warner Chilcott Investigational Study Site, Aventura, Florida
  - Warner Chilcott Investigational Study Site, Clearwater, Florida
  - Warner Chilcottt Investigational Study Site, Clearwater, Florida
  - Warner Chilcott Investigational Study Site, Hialeah, Florida
  - Warner Chilcott Investigational Study Site, Jacksonville, Florida
  - Warner Chilcott Investigational Study Site, Kissimmee, Florida
  - Warner Chilcott Investigational Study Site, Miami, Florida
  - Warner Chilcott Investigational Study Site, Ocala, Florida
  - Warner Chilcott Investigational Study Site, Pembroke Pines, Florida
  - Warner Chilcott Investigational Study Site, Tallahassee, Florida
  - Warner Chilcott Investigational Study Site, Atlanta, Georgia
  - Warner Chilcott Investigational Study Site, Sandy Springs, Georgia
  - Warner Chilcott Investigational Study Site, Coeur d'Alene, Idaho
  - Warner Chilcott Investigational Study Site, Chicago, Illinois
  - Warner Chilcott Investigational Study Site, Evanston, Illinois
  - Warner Chilcott Investigational Study Site, Melrose Park, Illinois
  - Warner Chilcott Investigational Study Site, Springfield, Illinois
  - Warner Chilcott Investigational Study Site, Anderson, Indiana
  - Warner Chilcott Investigational Study Site, Fort Wayne, Indiana
  - Warner Chilcott Investigational Study Site, Jeffersonville, Indiana
  - Warner Chilcott Investigational Study Site, Muncie, Indiana
  - Warner Chilcott Investigational Study Site, Newburgh, Indiana
  - Warner Chilcott Investigational Study Site, West Des Moines, Iowa
  - Warner Chilcott Investigational Study Site, Overland Park, Kansas
  - Warner Chilcott Investigational Study Site, Shreveport, Louisiana
  - Warner Chilcott Investigational Study Site, Elkridge, Maryland
  - Warner Chilcott Investigational Study Site, Glen Burnie, Maryland
  - Warner Chilcott Investigational Study Site, Owing Mills, Maryland
  - Warner Chilcott Investigational Study Site, Towson, Maryland
  - Warner Chilcott Investigational Study Site, Brookline, Massachusetts
  - Warner Chilcott Investigational Study Site, Omaha, Nebraska
  - Warner Chilcott Investigational Study Site, Las Vegas, Nevada
  - Warner Chilcott Investigational Study Site, Lawrenceville, New Jersey
  - Warner Chilcott Investigational Study Site, Albuquerque, New Mexico
  - Warner Chilcott Investigational Study Site, Albany, New York
  - Warner Chilcott Investigational Study Site, Brooklyn, New York
  - Warner Chilcott Investigational Study Site, Garden City, New York
  - Warner Chilcott Investigational Study Site, Great Neck, New York
  - Warner Chilcott Investigational Study Site, Kingston, New York
  - Warner Chilcott Investigational Study Site, New York, New York
  - Warner Chilcott Investigational Study Site, Newburgh, New York
  - Warner Chilcott Investigational Study Site, Poughkeepsie, New York
  - Warner Chilcott Investigational Study Site, Cary, North Carolina
  - Warner Chilcott Investigational Study Site, Charlotte, North Carolina
  - Warner Chilcott Investigational Study Site, Concord, North Carolina
  - Warner Chilcott Investigational Study Site, High Point, North Carolina
  - Warner Chilcott Investigational Study Site, Raleigh, North Carolina
  - Warner Chilcott Investigational Study Site, Salisbury, North Carolina
  - Warner Chilcott Investigational Study Site, Wilmington, North Carolina
  - Warner Chilcott Investigational Study Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Study Site, Cincinnati, Ohio
  - Warner Chilcott Investigational Study Site, Columbus, Ohio
  - Warner Chilcott Investigational Study Site, Lyndhurst, Ohio
  - Warner Chilcott Investigational Study Site, Bala-Cynwyd, Pennsylvania
  - Warner Chilcott Investigational Study Site, Lancaster, Pennsylvania
  - Warner Chilcott Investigational Study Site, Reading, Pennsylvania
  - Warner Chilcott Investigational Study Site, Warwick, Rhode Island
  - Warner Chilcott Investigational Study Site, Charleston, South Carolina
  - Warner Chilcott Investigational Study Site, Myrtle Beach, South Carolina
  - Warner Chilcott Investigational Study Site, Bristol, Tennessee
  - Warner Chilcott Investigational Study Site, Austin, Texas
  - Warner Chilcott Investigational Study Site, Dallas, Texas
  - Warner Chilcott Investigational Study Site, San Antonio, Texas
  - Warner Chilcott Investigational Study Site, Salt Lake City, Utah
  - Warner Chilcott Investigational Study Site, Virginia Beach, Virginia
  - Warner Chilcott Investigational Study Site, Winchester, Virginia
  - Warner Chilcott Investigational Study Site, Mountlake Terrace, Washington
  - Warner Chilcott Investigational Study Site, Wauwatosa, Wisconsin